CLINICAL TRIAL: NCT02561364
Title: Pattern of Human Fetal Biophysical Profile Scoring in Relationship to Gestational Age.
Brief Title: Biophysical Profile in Preterm Pregnancies
Acronym: BPP
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 15-03853-XP
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2016-10

CONDITIONS: Fetal Development
Keywords: Fetal Biophysical Profile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the fetal biophysical profile (BPP) scoring in pregnant women from 20 weeks-0 days' to 36 weeks-6 days' gestation. A biophysical profile (BPP) is a score that is intended to assess fetal well-being. This test will be performed within the expected time of the routine ultrasound exam.

DETAILED DESCRIPTION:
1. PURPOSE: To determine whether human fetal biophysical profile (BPP) scoring varies according to gestational age in preterm pregnancies.
2. RATIONALE: Fetal BPP and non-stress tests (NST) are useful tools in the assessment of fetal well-being in term fetuses. While for NST it has been established that the criteria for reassuring well-being are less strict in premature fetuses below 32 weeks' gestation, the pattern of BPP scoring according to preterm gestational age has not been fully investigated. The investigators consider that in premature fetuses, a reassuring BPP scoring does not need to be as strict as that used in term fetuses.
3. STUDY/PROJECT POPULATION:

   The Investigators' aim to use BPP scoring during routine ultrasound visits that pregnant patients undergo as part of their prenatal care. A routine ultrasound visit is performed during 30 to 60 minutes. The use of BPP will not add additional time to that taken by the routine ultrasound visit.

   The investigators will use BPP scoring in women from 20 to 36 weeks' gestation who attend routine ultrasound visits at the MedPlex Outpatient Clinic - Regional One Health. The sonographers are trained in the performance of BPP. The investigators will include women with singleton and multiple pregnancies who are able to provide informed consent.

   The investigators will exclude women who do not consent for the study, those unable to provide informed consent, and those with lethal fetal anomalies.
4. RESEARCH DESIGN Descriptive study with prospective collection of data.
5. STUDY/PROJECT PROCEDURES:

   The study will involve the performance of a biophysical profile (BPP) scoring during routine ultrasound exams. The BPP is not intended to last more than 30 minutes. A BPP score is composed by ultrasound assessment of:
   * amniotic fluid volume (normal = 2 points, low = 0 points)
   * fetal movements (3 or more movements = 2 points, less movements = 0 points); we will record the total number of movements during the testing period
   * fetal breathing (sustained 30 second breathing = 2 points, <30 seconds = 0 points); we will record time of sustained breathing during the testing period
   * fetal tone (extension and flexion = 2 points, lack of extension/flexion = 0 points) For those patients undergoing standard of care scheduled BPP, information will be abstracted from the scheduled test.

   For those patients undergoing standard of care ultrasound but are not scheduled for BPP, additional BPP will be obtained within the time allotted for the already scheduled ultrasound.

   The investigators will correlate the BPP scoring with the non-stress test (NST) or Doppler flow reports in those fetuses already undergoing NST or Doppler studies for other obstetric indications not related to the purpose of this study.
6. OUTCOME MEASURES:

Primary outcome: fetal or neonatal survival

Secondary outcomes:

* gestational age at delivery
* need for NST
* hospitalization
* need for antenatal steroids use
* fetal growth restriction
* spontaneous or indicated preterm delivery
* neonate apgars
* neonatal morbidity: respiratory, gastrointestinal, neurologic, metabolic

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 20 wks 0 days and 36 wks and 6 days
* singleton or multiple pregnancies
* able to provide informed consent
* age 18 to 45 years old

Exclusion Criteria:

* lethal fatal anomalies
* those not providing informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant patients that meet the all of the inclusion criteria and do not meet the exclusion criteria, will be approached during their routine prenatal care regarding their interest in participation. Women must be between 20 weeks to 36 weeks of their pregnancy.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Fetal or neonatal survival measured as live birth or fetal demise | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants

SECONDARY OUTCOMES:
gestational age at delivery as measured by ultrasound calculations | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
need for non-stress test as necessary for related health issue, determined by the health history and measured by occurrence with supporting health documentation | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
hospitalization measured as necessary for related health issue with documentation of procedures and length of stay | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
need for antenatal steroids use as indicated for high risk of preterm delivery measured as necessary for related health issue, and utilized. | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
fetal growth restriction (FGR) measured by American College of Obstetricians and Gynecologists (ACOG): FGR: Fetus-estimated weight below 10th percentile. small for gestational age (SGA): Newborns-weight below the 10th percentile for gestational age. | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
spontaneous or indicated preterm delivery documented as occurring or necessary for related health issue | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
neonate apgar scores measured at birth: At 1 minute and 5 minutes (scoring 0, 1,or 2 in 5 physiological functions: Activity (muscle tone), Pulse (heart rate), Grimace (reflex response), Appearance (color), and Respiration (breathing)]. | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants
Number of neonates born with morbid conditions: respiratory, gastrointestinal, neurologic, metabolic; documented as present. | 20 weeks 0 days up to 36 weeks and 6 days
  will be monitored and recorded on all participants

CONTACTS AND LOCATIONS:
Overall Officials: Luis M. Gomez, M.D., Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Regional One Health Ob-Gyn Clinic, Memphis, Tennessee
  - Regional One Health Center for High Risk Pregnancies, Memphis, Tennessee

REFERENCES:
- [Background] Harman, CR. Assessment of Fetal Health. In: Creasy RK, Resnik R, Iams JD, Lockwood CJ, Moor TM, editors. Maternal-fetal medicine: principle and practice. 6th ed. Philadelphia (PA):Saunders 2009. p. 361-95.
- [Background] American College of Obstetricians and Gynecologists. Practice bulletin no. 116: Management of intrapartum fetal heart rate tracings. Obstet Gynecol. 2010 Nov;116(5):1232-40. doi: 10.1097/AOG.0b013e3182004fa9. PMID 20966730
- [Background] Macones GA, Hankins GD, Spong CY, Hauth J, Moore T. The 2008 National Institute of Child Health and Human Development workshop report on electronic fetal monitoring: update on definitions, interpretation, and research guidelines. Obstet Gynecol. 2008 Sep;112(3):661-6. doi: 10.1097/AOG.0b013e3181841395. PMID 18757666
- [Background] Druzin ML, Smith JF, Gabbe SG, Reed KL, Antepartum Fetal Evaluation. In: Gabbe SG, Niebyl JR Simpson JL, editors. Obstetrics: normal and problem pregnancies. 5th ed. Philadelphia (PA): Churchill Livingstone; 2007. p. 267-300.
- [Result] Druzin ML, Fox A, Kogut E, Carlson C. The relationship of the nonstress test to gestational age. Am J Obstet Gynecol. 1985 Oct 15;153(4):386-9. doi: 10.1016/0002-9378(85)90075-4. PMID 3901768
- [Result] Gagnon R, Campbell K, Hunse C, Patrick J. Patterns of human fetal heart rate accelerations from 26 weeks to term. Am J Obstet Gynecol. 1987 Sep;157(3):743-8. doi: 10.1016/s0002-9378(87)80042-x. PMID 3631176
- [Result] Natale R, Nasello C, Turliuk R. The relationship between movements and accelerations in fetal heart rate at twenty-four to thirty-two weeks' gestation. Am J Obstet Gynecol. 1984 Mar 1;148(5):591-5. doi: 10.1016/0002-9378(84)90754-3. PMID 6702921
- [Result] Sorokin Y, Dierker LJ, Pillay SK, Zador IE, Schreiner ML, Rosen MG. The association between fetal heart rate patterns and fetal movements in pregnancies between 20 and 30 weeks' gestation. Am J Obstet Gynecol. 1982 Jun 1;143(3):243-9. doi: 10.1016/0002-9378(82)90812-2. PMID 7081342
- [Result] Baskett TF. Gestational age and fetal biophysical assessment. Am J Obstet Gynecol. 1988 Feb;158(2):332-4. doi: 10.1016/0002-9378(88)90149-4. PMID 3341411